CLINICAL TRIAL: NCT02224625
Title: Randomized and Observer-blinded Study to Evaluate the Cumulative Irritation and Contact Sensitizing Potential of One Finished Test Product
Brief Title: Irritation and Sensitization of Chlorhexidine Gluconate (CHG) Cloth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R13-051
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2016-03

CONDITIONS: Surgery
MeSH Terms: interventions — chlorhexidine gluconate; Sodium Chloride; Sodium Dodecyl Sulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2% CHG Cloth (Experimental): Chlorhexidine Gluconate 2%
  Interventions: Drug: 2% CHG Cloth solution
- Vehicle Cloth (Placebo Comparator): Excipients on cloth
  Interventions: Device: Vehicle Cloth
- DynaHex (2% CHG) (Active Comparator): Chlorhexidine Gluconate 2% solution
  Interventions: Drug: Active Comparator
- Saline (Sham Comparator): 0.9% sodium chloride
  Interventions: Other: Saline
- Sodium Lauryl Sulfate (SLS) (Active Comparator): Sodium lauryl sulfate to produce mild irritation as a positive control
  Interventions: Other: SLS

INTERVENTIONS:
Drug: 2% CHG Cloth solution — Investigational CHG
  Other Names: Chlorhexidine Gluconate
  Arms: 2% CHG Cloth
Device: Vehicle Cloth — Excipients from CHG cloth only
  Other Names: Control
  Arms: Vehicle Cloth
Drug: Active Comparator — Active comparator
  Other Names: DynaHex-2
  Arms: DynaHex (2% CHG)
Other: Saline — Negative control
  Arms: Saline
Other: SLS — Provides a slight irritation for a positive control
  Other Names: Sodium Lauryl Sulfate
  Arms: Sodium Lauryl Sulfate (SLS)

SUMMARY:
Evaluating the irritation properties of CHG cloth. Some Subjects will also have the product applied to see if they become sensitized to repeated applications.

DETAILED DESCRIPTION:
For the Irritation Study (30 subjects), patches containing CHG, vehicle, saline, CHG comparator or sodium lauryl sulfate (a product that is expected to produce a slight skin irritation) will be placed on the same spot of your skin every day for 21 days. The skin will be examined every day.

The Sensitization Study (200 total subjects) place patches containing CHG, vehicle, saline, CHG comparator on the skin 3 times a week for 3 weeks. Following a two-week rest period the patches will be reapplied for 48 hours and assessed out to 72 hours thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Free of skin disorders
* Signed consent

Exclusion Criteria:

* Allergies to latex
* Topical or systemic steroids, antihistamines, antiinflammatory agents 7 days prior or during testing
* severe illness
* Pregnant (females)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Pullman, MD, Principal Investigator — BioScience Laboratories
Locations (1):
- BioScience Laboratories, Butte, Montana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared with FDA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 of the 249 participants participated in both the Irritation and Sensitization Studies.
Pre-assignment Details: Participants received up to 5 products simultaneously on their skin. SLS was only used in the Irritation study (39 subjects) as a positive control.
Groups:
- 2% CHG Cloth, Vehicle, DynaHex, Saline, SLS: Chlorhexidine Gluconate 2% cloth solution Vehicle solution of 2% CHG cloth DynaHex (2% CHG) 0.9% Saline Sodium Lauryl Sulfate
Period: Irritation
Arm/Group | 2% CHG Cloth, Vehicle, DynaHex, Saline, SLS
Started | 39
Completed | 33
Not Completed | 6
Not completed — Adverse Event | 6
Period: Sensitization
Arm/Group | 2% CHG Cloth, Vehicle, DynaHex, Saline, SLS
Started | 249 (Subjects from Irritation study also participated in Sensitization Study)
Completed | 194
Not Completed | 55
Not completed — Adverse Event | 55

BASELINE CHARACTERISTICS:
Population: Participants in the Sensitization study received the following 4 products ( 2% CHG cloth, Vehicle cloth, DynaHex and Saline). Participants in the Irritation study received the same 4 products in addition to SLS.
Groups:
- 2% CHG, Vehicle, DynaHex, Saline: Chlorhexidine Gluconate 2% Cloth Solution Vehicle solution of CHG cloth DynaHex 2% CHG solution 0.9% Saline Sodium Lauryl Sulfate (only used in Irritation Study)
Arm/Group | 2% CHG, Vehicle, DynaHex, Saline
Number analyzed (Participants) | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 226
  >=65 years | 15
Age, Continuous [Mean (Full Range); unit: years] | 38 [16 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 102
Region of Enrollment [Number; unit: participants]
  United States | 249

OUTCOME MEASURES:

1. Primary Outcome: Grading Scale for Visual Evaluation of Skin Condition
Description: Irritation: 21 days of patching (total). A reviewer will assign a score based on an 8 point categorical scale to the areas treated at each visit.
  Sensitization: 35 days (21 days of patching followed by 14 days rest and subsequent patch). A reviewer will assign a score based on an 8 point categorical scale to the areas treated at each visit. SLS was not tested.
  Grade 0 = No irritation Grade 1 = Minimal erythema Grade 2 = Definite erythema Grade 3 = Erythema and papules Grade 4 = Edema Grade 5 = Erythema, edema and papules Grade 6 = Vesicular eruption Grade 7 = Strong reaction spreading
Time Frame: 21 Days for Irritation (N=39). 35 Days for Sensitization (N=249)
Population: Participants received more than one product at a time.
Measure: Mean (Full Range); unit: Scores Ranging (0-7)
Groups:
- 2% CHG Cloth: Chlorhexidine Gluconate 2%
  2% CHG Cloth: CHG solution on cloth
- DynaHex (2% CHG): Chlorhexidine Gluconate 2% solution
  Active Comparator: 2% CHG solution
Arm/Group | 2% CHG Cloth | Vehicle Cloth | DynaHex (2% CHG) | Saline | Sodium Lauryl Sulfate (SLS)
Number analyzed (Participants) | 249 | 249 | 249 | 249 | 39
Scores Ranging (0-7)
  Irritation Mean Visualization Score Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Irritation Mean Visualization Score Day 21 | 2.9 [0 to 4] | 1.4 [0 to 4] | 3.3 [3 to 4] | 0.7 [0 to 3] | 3.0 [3 to 3]
  Sensitization Mean Visualization Score Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Sensitization Mean Visualization Score Day 35 | 0.12 [0 to 2] | 0.03 [0 to 2] | 0.03 [0 to 2] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events reported over a 21 (irritation) and 35 (sensitization) day period.
Description: Participants received up to 5 different products simultaneously during the study. Adverse skin reactions with known relationships to the products applied were reported individually. Non-skin related adverse events were also captured during the study but could not be associated directly with a particular treatment and are not included.
Arm/Group | 2% CHG Cloth | Vehicle Cloth | DynaHex (2% CHG) | Saline | Sodium Lauryl Sulfate (SLS)
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/249 | 0/249 | 0/249 | 0/39
Other Adverse Events (participants affected / at risk) | 5/249 | 0/249 | 15/249 | 0/249 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2% CHG Cloth (N=249) | Vehicle Cloth (N=249) | DynaHex (2% CHG) (N=249) | Saline (N=249) | Sodium Lauryl Sulfate (SLS) (N=39)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 12 (12) | 0 (0) | 0 (0)
Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential information based on contract